CLINICAL TRIAL: NCT02598739
Title: Resistance Training in Patients With Psoriatic Arthritis Improves Function, Disease Activity and Quality of Life
Brief Title: Evaluation of the Effectiveness of Resistance Training in Patients With Psoriatic Arthritis
Acronym: PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Diego Roger Silva, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0196/11
Record Dates: First submitted 2014-08-19; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Psoriatic Arthritis
Keywords: Physical exercise; Psoriatic arthritis; Quality of life
MeSH Terms: conditions — Arthritis, Psoriatic; Motor Activity | interventions — Resistance Training; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance exercise (Experimental): Underwent resistance exercise twice a week, for twelve weeks for the following muscles group: upper limbs, lower limbs and trunk.
  It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises were 60% of one-maximum repetition (1RM).
  The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteo: standing hips extension.
  Interventions: Other: Resistance exercise
- Control group (Other): Waiting list for the exercises.
  Interventions: Other: Waiting list for the exercises

INTERVENTIONS:
Other: Resistance exercise — Underwent resistance exercise twice a week, for twelve weeks. The IG patients performed resistance exercises for the following muscles group: upper limbs, lower limbs and trunk.
  It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises were 60% of one-maximum repetition (1RM).
  The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteo: standing hips extension.
  Arms: Resistance exercise
Other: Waiting list for the exercises
  Arms: Control group

SUMMARY:
The aim of this study was to assess the effectiveness of resistance training in improving functional capacity, muscle strength, quality of life and disease activity in patients with PSA.

DETAILED DESCRIPTION:
The IG patients performed resistance exercises for the following muscles group: upper limbs, lower limbs and trunk. It was used a machine "leg extension" for the training on the lower limbs. For upper limbs we used a pulley triceps machine and front pull in addition to free weights (dumbbells).

In order to perform the exercise program the study followed all the recommendations established by the American College of Sports Medicine (ACSM) (Ratamess et al., 2009). It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises were 60% of one-maximum repetition (1RM).

The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteo: standing hips extension.

Control Group (CG) The control group was kept in a waiting list while continued with the standard pharmacological treatment during all the study. The patients were instructed to maintain their daily activities and to avoid any other non-pharmacological treatment. The exercise program was offered to the control group in the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of psoriatic arthritis, according to the CASPAR criteria
* Between 18 and 65 years of age, of both genders who agreed and signed the consent form.
* Patients should be-modifying drugs (DMARDs) on stable doses for at least three months and doses of non-steroidal anti-inflammatory drugs and corticosteroids stable for at least 4 weeks

Exclusion Criteria:

Patients were excluded:

* Uncontrolled cardiovascular disease
* Decompensated diabetes mellitus; diseases
* Severe psychiatric
* Fibromyalgia
* Other medical conditions that most disabling EA
* History of regular exercise (at least 30 minutes 2 times per week) during the last 6 months
* Arthroplasties of the hip and / or knee in the last 12 months; AND
* Any other medical condition that prevents the patient from performing resistance exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the functional capacity | Baseline, after 45 and 90 days
  Evaluated by HAQ-S Health Assessment Questionnaire for the Spondylarthropathies

SECONDARY OUTCOMES:
Change in the quality of life | Baseline, after 45 and 90 days
  Evaluated by the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PHD, Study Chair — Federal University of São Paulo
Locations (1):
- São Paulo Hospital, São Paulo, São Paulo, Brazil